CLINICAL TRIAL: NCT01741454
Title: Combination Versus Monotherapy With Alpha Blocker and Anticholinergics to Relieve Urinary Stent Symptoms
Brief Title: Treatment of Symptoms After Stent Placement for Urinary Tract Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-0755; 2012-0279 (Other: HS IRB)
Record Dates: First submitted 2012-11-29; First posted 2012-12-05 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Ureteral Obstruction
Keywords: Tolterodine; Tamsulosin; Ureteral Obstruction
MeSH Terms: conditions — Ureteral Obstruction | interventions — Tamsulosin; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tamsulosin plus placebo 7-day treatment (Active Comparator): Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Interventions: Drug: Tamsulosin
- Tamsulosin plus Tolterodine ER 7-day treatment (Experimental): Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Interventions: Drug: Tamsulosin; Drug: Tolterodine ER
- Tamsulosin plus placebo 21-day treamtnet (Active Comparator): Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Interventions: Drug: Tamsulosin
- Tamsulosin plus Tolterodine ER 21-day treatment (Experimental): Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Interventions: Drug: Tamsulosin; Drug: Tolterodine ER

INTERVENTIONS:
Drug: Tamsulosin — 0.4 mg by mouth once per day.
  Other Names: Flomax (TM)
Drug: Tolterodine ER — 4 mg by mouth once a day.
  Other Names: Detrol (TM)
  Arms: Tamsulosin plus Tolterodine ER 21-day treatment; Tamsulosin plus Tolterodine ER 7-day treatment

SUMMARY:
The purpose of this study is to determine whether combination therapy with Tolterodine ER and Tamsulosin is more effective than monotherapy with tamsulosin alone in reducing stent symptoms. The second purpose is to determine if people have less stent discomfort if they take these medications starting 2 weeks before the stent is placed

The investigators hope to show that the addition of Tolterodine ER to Tamsulosin will provide added benefits in reducing stent symptoms in patients who have had unilateral placement of a ureteral stent.

DETAILED DESCRIPTION:
The investigators aim to show that the addition of Tolterodine ER to Tamsulosin will provide added benefits in ameliorating stent-related symptoms in participants who have had unilateral placement of a ureteral stent for urolithiasis. This objective will be assessed by determining the mean difference in the urinary symptom index domain of the Urinary Stent Symptom Questionnaire, which is a validated tool used to assess stent symptoms. The investigators suggest that a 15% further decrease in the index score in the experimental group, compared to the control group would represent a clinically significant improvement in urinary symptoms, based on the prior studies evaluating lower urinary tract symptoms in patients with stents. The investigators hypothesize that combination therapy with Tamsulosin and Tolterodine ER will yield greater symptom relief than tamsulosin alone.

Initially, a 7-day design (medical starts 7 days before stent insertion) was conducted to determine whether combination therapy with Tolterodine ER and Tamsulosin is more effective than monotherapy with tamsulosin alone in reducing stent symptoms.

Previous studies showed that tolterodine ER therapy significantly reduces urinary symptoms by week 4 of medication therapy. Given the evidence that tolterodine ER requires a longer duration to have maximum benefit, in the second phase, investigators increased the duration of medication to start 2 weeks prior to surgery and continued for 7 days after surgery, for a total of 21 days of medication, to test whether combination therapy is more effective than monotherapy in reducing stent symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral ureteral stent placement for urolithiasis

Exclusion Criteria:

1. Pre-existing lower urinary tract symptoms
2. Active urinary tract infection
3. Contraindication to anticholinergic medication

   1. Prior hypersensitivity or allergy to tolterodine
   2. Patients with severe hepatic impairment (Child-Pugh Class C)
   3. Patients with uncontrolled close (narrow) angle glaucoma
   4. Patients with urinary retention
4. Current anticholinergic use
5. Chronic pelvic pain syndromes (e.g. acute/chronic prostatitis, interstitial cystitis)
6. Women who are pregnant or nursing
7. Under 18 years of age
8. Prior hypersensitivity or allergy to tolterodine
9. Patients with severe hepatic impairment (Child-Pugh Class C)
10. Patients with uncontrolled close (narrow) angle glaucoma
11. Patients with urinary retention
12. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2012-11; Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nakada, MD, Principal Investigator — Univeristy of Wisconsin
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment is slow, drop out rate is high, thus, we decide to stop enrolling.
Groups:
- Tamsulosin Plus Placebo 7 Day: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tamsulosin: 0.4 mg by mouth once per day for 7 days
- Tamsulosin Plus Tolterodine ER 7 Day: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Tamsulosin: 0.4 mg by mouth once per day for 7 days
  Tolterodine ER: 4 mg by mouth once a day for 7 days
- Tamsulosin Plus Placebo 21 Day: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tamsulosin: 0.4 mg by mouth once per day for 21 days
- Tamsulosin Plus Tolterodine ER 21 Day: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Tamsulosin: 0.4 mg by mouth once per day for 21 days
  Tolterodine ER: 4 mg by mouth once a day for 21 days
Period: Overall Study
Arm/Group | Tamsulosin Plus Placebo 7 Day | Tamsulosin Plus Tolterodine ER 7 Day | Tamsulosin Plus Placebo 21 Day | Tamsulosin Plus Tolterodine ER 21 Day
Started | 49 | 50 | 39 | 43
Completed | 36 | 44 | 22 | 21
Not Completed | 13 | 6 | 17 | 22

BASELINE CHARACTERISTICS:
Population: Patients who dropped out were not analyzed
Groups:
- Tamsulosin Plus Placebo 7 Day Treatment; Tamsulosin Plus Placebo 21 Day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tamsulosin: 0.4 mg by mouth once per day.
- Tamsulosin Plus Tolterodine ER 7 Day Treatment; Tamsulosin Plus Tolterodine ER 21 Day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Tamsulosin: 0.4 mg by mouth once per day.
  Tolterodine ER: 4 mg by mouth once a day.
- Total: Total of all reporting groups
Arm/Group | Tamsulosin Plus Placebo 7 Day Treatment | Tamsulosin Plus Tolterodine ER 7 Day Treatment | Tamsulosin Plus Placebo 21 Day Treatment | Tamsulosin Plus Tolterodine ER 21 Day Treatment | Total
Number analyzed (Participants) | 36 | 44 | 22 | 21 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (18) | 51.5 (12.7) | 57.3 (10.3) | 56.9 (16.2) | 53.4 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 25 | 10 | 11 | 61
  Male | 21 | 19 | 12 | 10 | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 44 | 22 | 21 | 123

OUTCOME MEASURES:

1. Primary Outcome: Ureteral Stent Symptom Questionnaire Score Up to 24 Hours Prior to Stent Insertion
Description: The ureteral stent symptom questionnaire contains 36 items from the 5 subscales: urinary index (11-items, total range of scores 11-54, The range of the mean score is 1-4.9), pain (8-items, total range of scores 5-27. Two items are not included in the calculation. The range of the mean score is 0.83-4.5), general health (6-items, total range of scores 4-28. The range of the mean score is 0.67-4.67), work (if stent influence patients work; 7-items, total range of scores 3-15. Four items are not included in the calculation. The range of the mean score is 1-5), and sexual matters (4-items, total range of scores 2-10. Two items are not included in the calculation. The range of the mean score is 1-5). In all cases, higher scores indicate worse outcomes. The score for each subscale is summed and divided by the number of items on the subscale. The group mean for each subscale is reported, the score is not normalized.
Time Frame: Up to 24 hours prior to stent insertion
Population: For all sub-scales, we reported the average score, the higher values suggest worse outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tamsulosin Plus Placebo 7-day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tamsulosin: 0.4 mg by mouth once per day for 7 dyas
- Tamsulosin Plus Tolterodine ER 7-day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Tamsulosin: 0.4 mg by mouth once per day for 7 days
  Tolterodine ER: 4 mg by mouth once a day for 7 days
- Tamsulosin Plus Placebo 21-day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tamsulosin: 0.4 mg by mouth once per day for 21 dyas
- Tamsulosin Plus Tolterodine ER 21-day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Tamsulosin: 0.4 mg by mouth once per day for 21days
  Tolterodine ER: 4 mg by mouth once a day for 21 days
Arm/Group | Tamsulosin Plus Placebo 7-day Treatment | Tamsulosin Plus Tolterodine ER 7-day Treatment | Tamsulosin Plus Placebo 21-day Treatment | Tamsulosin Plus Tolterodine ER 21-day Treatment
Number analyzed (Participants) | 36 | 44 | 22 | 21
score on a scale
  Urinary index | 1.76 (0.46) | 1.84 (0.39) | 2.02 (0.27) | 1.93 (0.48)
  Pain score | 1.95 (0.74) | 2.13 (0.94) | 2.49 (0.7) | 1.88 (0.7)
  General health score | 1.87 (0.55) | 2.04 (0.83) | 2.15 (0.6) | 2.07 (0.6)
  Work | 1.65 (0.83) | 1.76 (0.91) | 2.05 (0.96) | 1.18 (0.4)
  Sexual matters | 1.60 (0.6) | 1.41 (0.41) | 1.77 (0.73) | 1.57 (0.63)

2. Primary Outcome: Ureteral Stent Symptom Questionnaire Score
Description: as for outcome 1
Time Frame: 42-48 hours post-stent insertion
Population: Same
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tamsulosin Plus Tolterodine ER 7-day Treatment; Tamsulosin Plus Tolterodine ER 21-day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tolterodine ER is an anticholinergic agent, which is used as one of the first line agents for detrusor overactivity.
  Tamsulosin: 0.4 mg by mouth once per day.
  Tolterodine ER: 4 mg by mouth once a day.
- Tamsulosin Plus Placebo 21-day Treatment: Tamsulosin is a selective α1a-blocker (FlomaxTM), generic since 2009. It is an antagonist of α1-mediated contraction of prostate, bladder and proximal urethral smooth muscle, and as such, reduces urethral pressure and resistance, bladder outlet resistance, bladder hyperactivity, and consequently lower urinary tract symptoms.
  Tamsulosin: 0.4 mg by mouth once per day.
Arm/Group | Tamsulosin Plus Placebo 7-day Treatment | Tamsulosin Plus Tolterodine ER 7-day Treatment | Tamsulosin Plus Placebo 21-day Treatment | Tamsulosin Plus Tolterodine ER 21-day Treatment
Number analyzed (Participants) | 36 | 44 | 22 | 21
score on a scale
  Urinary index | 2.95 (0.45) | 2.91 (0.55) | 2.98 (0.64) | 2.83 (0.63)
  Pain score | 2.66 (0.79) | 2.89 (0.98) | 2.9 (0.95) | 2.71 (0.76)
  General health score | 2.35 (0.74) | 2.69 (0.85) | 2.64 (0.85) | 2.78 (0.95)
  Work | 2.04 (0.97) | 2.92 (1.29) | 2.1 (1.05) | 1.79 (1.21)
  Sexual matters | 2.07 (1.01) | 2 (0.91) | 1.83 (0.76) | 1.75 (1.06)

3. Primary Outcome: Ureteral Stent Symptom Questionnaire Score 5-7 Days Post-stent Insertion
Description: as for outcome 1
Time Frame: 5-7 days post-stent insertion
Population: same
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tamsulosin Plus Placebo 7-day Treatment | Tamsulosin Plus Tolterodine ER 7-day Treatment | Tamsulosin Plus Placebo 21-day Treatment | Tamsulosin Plus Tolterodine ER 21-day Treatment
Number analyzed (Participants) | 36 | 44 | 22 | 21
score on a scale
  Urinary index | 2.46 (0.58) | 2.55 (0.63) | 2.49 (0.48) | 2.46 (0.66)
  Pain score | 2.39 (0.94) | 2.49 (0.97) | 2.58 (0.83) | 2.4 (0.86)
  General health score | 2.34 (0.92) | 2.33 (0.8) | 2.52 (0.83) | 2.28 (0.75)
  Work | 2.81 (0.88) | 2.61 (1.19) | 1.94 (1.05) | 1.47 (0.67)
  Sexual matters | 1.5 (0.4) | 1.59 (0.76) | 1.75 (0.69) | 2.9 (1.19)

4. Primary Outcome: Ureteral Stent Symptom Questionnaire Score Up to 24 Hours After Stent Removal
Description: as for outcome 1
Time Frame: Up to 24 hours after stent removal. Removal will occur 5 to 7 days after insertion.
Population: same
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tamsulosin Plus Placebo 7-day Treatment | Tamsulosin Plus Tolterodine ER 7-day Treatment | Tamsulosin Plus Placebo 21-day Treatment | Tamsulosin Plus Tolterodine ER 21-day Treatment
Number analyzed (Participants) | 36 | 44 | 22 | 21
score on a scale
  Urinary index | 1.72 (0.45) | 1.91 (0.53) | 1.85 (0.46) | 2.14 (0.61)
  Pain score | 1.66 (0.91) | 1.66 (0.79) | 1.97 (1.01) | 2.08 (0.47)
  General health score | 1.73 (0.71) | 1.67 (0.62) | 1.84 (1.02) | 1.99 (0.75)
  Work | 1.57 (0.95) | 1.41 (0.57) | 2.13 (1.36) | 1.56 (0.91)
  Sexual matters | 1.42 (0.4) | 1.3 (0.35) | 1.58 (0.58) | 2.42 (1.5)

ADVERSE EVENTS:
Time Frame: from the first week of enrollment to 6 months.
Description: The study drugs being used are Tamsulosin and Tolterodine ER. Both drugs are FDA-approved for treating specific conditions and are routinely used in urology for other conditions as well. Previous studies showed that most of side effects are bothersome at worst to the patient.
Arm/Group | Tamsulosin Plus Placebo 7 Day Treatment | Tamsulosin Plus Tolterodine ER 7 Day Treatment | Tamsulosin Plus Placebo 21 Day Treatment | Tamsulosin Plus Tolterodine ER 21 Day Treatment
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50 | 0/39 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50 | 0/39 | 0/43
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50 | 0/39 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT01741454/Prot_SAP_000.pdf